CLINICAL TRIAL: NCT07204457
Title: Multicenter, Randomized, Subject/Evaluator Blind, Active Control, Phase II/III Clinical Trial to Assess Immunogenicity and Safety of EG-MCV4 Meningococcal (Groups A, C, W-135, and Y) Conjugated Vaccines
Brief Title: Immunogenicity and Safety of Meningococcal Conjugate Vaccine (EG-MCV4) in Healthy Adults Aged 19 to 55 Years Old
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: EyeGene Inc. (Other)
Collaborators: BMI Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EG-MCV4-P3
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Meningococcal Infections
Keywords: Meningococcal Vaccines; Vaccines, Conjugate; Bacterial Vaccines; Vaccines; Bacterial Infections; Meningococcal Disease; Neiseriaceae Infections; Gram-Negative Bacterial Infections; Infections; Biological Products
MeSH Terms: conditions — Meningococcal Infections; Bacterial Infections; Gram-Negative Bacterial Infections; Infections | interventions — Vaccines, Conjugate; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EG-MCV4 (Test group 1) (Experimental): Healthy adults received 0.5 mL single intramuscular dose on Day 0.
  Interventions: Biological: EG-MCV4
- EG-MCV4 (Test group 2) (Experimental): Healthy adults received 0.25 mL single intramuscular dose on Day 0.
  Interventions: Biological: EG-MCV4
- Menveo (Active Comparator): Healthy adults received 0.5 mL single intramuscular dose on Day 0.
  Interventions: Biological: Menveo

INTERVENTIONS:
Biological: EG-MCV4 — single intramuscular dose on Day 0
  Other Names: Meningococcal(Groups A, C, W-135, and Y) Conjugate Vaccine
  Arms: EG-MCV4 (Test group 1); EG-MCV4 (Test group 2)
Biological: Menveo — single intramuscular dose on Day 0
  Other Names: Meningococcal(Groups A, C, W-135, and Y) Conjugate Vaccine
  Arms: Menveo

SUMMARY:
Phase 2/3 study to evaluate immunogenicity and safety in healthy adult participants following a single dose administration of Meningococcal (groups A, C, W-135, and Y) conjugate vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 19 to 55 years.
* Individuals who have been fully informed about the clinical trial, understand the details, and voluntarily agree to participate by providing written informed consent.
* Individuals who are available for all scheduled visits, including phone calls and in-person appointments, for the duration of the study.

Exclusion Criteria:

* History of prior disease caused by N. meningitidis.
* Contact with a person infected with N. meningitidis within 60 days of screening.
* Prior receipt of a meningococcal vaccine or a vaccine containing a meningococcal antigen.
* History of or planned vaccination with any other vaccine within 4 weeks before or after administration of the investigational product.
* History of fever (≥ 38°C) within 3 days of screening, or a history of a significant acute infectious disease within 7 days of screening, or a chronic infectious disease within 4 weeks of screening.
* History of Hepatitis B or C at the time of screening.
* Presence of any significant acute, chronic, or progressive disease that, in the opinion of the investigator, could interfere with the conduct or completion of the study.
* History of malignancy or high-risk malignant disease within 5 years before the investigational product administration.
* History of epilepsy, progressive neurological disease, or Guillain-Barré Syndrome.
* History of anaphylaxis.
* History of systemic urticaria within 5 years of the investigational product administration.
* Hypersensitivity to the active substance, diphtheria toxoid (CRM197), or any other excipient, or a history of a life-threatening reaction to a vaccine containing similar components.
* Hypersensitivity to the investigational vaccine, any of its components, or latex.
* History of any therapy that could affect the immune system within 6 months of screening.
* History of immunodeficiency disease, or a family history of such a disease.
* Receipt of any parenteral immunoglobulin preparation, blood product, or plasma derivatives within 90 days of screening, or planned administration during the study period.
* History of platelet-related or hemorrhagic disorders or a history of excessive bleeding or bruising after intramuscular injection or venipuncture.
* Current treatment with anticoagulants or new antiplatelet agents.
* History of organ or bone marrow transplantation.
* Suspected history of drug or alcohol abuse within 1 year before the investigational product administration.
* Individuals unwilling to use a medically acceptable method of contraception for the duration of the clinical trial.
* Pregnant or lactating women.
* Receipt or planned receipt/application of another investigational drug or medical device within 6 months prior to study participation.
* Presence of a significant abnormality on a screening test, or any other reason that, in the opinion of the investigator, makes the individual unsuitable for the study.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1123 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Seroresponse | 28 days after the vaccination
  * Part 1:
    * The proportion of subjects achieving a seroresponse as measured by hSBA and rSBA
  * Part 2:
    * The proportion of subjects achieving a seroresponse as measured by rSBA

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Eunpyeong St.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No